CLINICAL TRIAL: NCT00062790
Title: Effects of Dutasteride on Intraprostatic Dihydrotestosterone (DHT) Levels
Brief Title: Effect Of Dutasteride On Intraprostatic Dihydrotestosterone (DHT) Levels
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ARI40014
Record Dates: First submitted 2003-06-16; First posted 2003-06-17 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Prostatic Hyperplasia
Keywords: Testosterone; DHT; TURP
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Dutasteride

INTERVENTIONS:
Drug: Dutasteride

SUMMARY:
This study is being done to determine how much certain hormone levels in the prostate decrease when a patient takes dutasteride 0.5mg daily for 3 months prior to TURP. Male patients at least 50 years old willing to take either dutasteride or a placebo (dummy pill) once daily by mouth for 3 months prior to having a surgery to reduce the size of their prostate. During the surgery, very small pieces of the prostate that are removed will be tested to see how much dihydrotestosterone and testosterone (male hormones) are in the tissue.

ELIGIBILITY:
Inclusion criteria:

* Diagnosed with benign prostatic hyperplasia
* Must be scheduled to have a transurethral resection of the prostate (prostate surgery) and be able to wait 3 months to have the procedure.
* PSA (prostate specific antigen) level must be between 1.5 and 15 ng/ml.

Exclusion criteria:

* Prostate cancer.
* Use of saw palmetto or other over the counter treatments for prostate health chemically related to the study medication.
* Previous finasteride use or other investigational 5ARI within 6 months prior to screening.
* History of chronic UTIs (urinary tract infections)
* Presence of acute bacterial prostatitis at screening

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2003-10; Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Effect of repeat oral daily dosing of 0.5mg dutasteride compared to placebo on prostate tissue content of DHT in patients treated for 3 months prior to transurethral resection of the prostate (TURP).

SECONDARY OUTCOMES:
Effect of repeat oral once daily dosing of 0.5mg dutasteride compared to placebo on prostatic tissue content of testosterone.
Changes in serum DHT (dihydrotestosterone) and T (testosterone).

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (11):
- United States (11):
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, New Britain, Connecticut
  - GSK Investigational Site, Trumbull, Connecticut
  - GSK Investigational Site, Augusta, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Niles, Illinois
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Lebanon, New Hampshire
  - GSK Investigational Site, Eugene, Oregon
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: ARI40014 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: ARI40014 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: ARI40014 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: ARI40014 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: ARI40014 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: ARI40014 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: ARI40014 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register